CLINICAL TRIAL: NCT00433771
Title: A Multi-Center, Single Arm, Prospective Study of the WallFlex™ Biliary Fully-covered Stent for the Palliative Treatment of Malignant Bile Duct Obstruction
Brief Title: A Study of the WallFlex™ Biliary Fully-covered Stent for the Palliative Treatment of Malignant Bile Duct Obstruction
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Jeremy Bolt, Boston Scientific
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ENDO-WALLFLEX-BIL-PALL-001U; E7009
Record Dates: First submitted 2007-02-08; First posted 2007-02-12 (Estimated); Results first posted 2010-02-09 (Estimated); Last update posted 2010-06-29 (Estimated); Status verified 2010-06

CONDITIONS: Cholestasis, Extrahepatic
Keywords: Malignant; Cholestasis, Extrahepatic; Biliary obstruction
MeSH Terms: conditions — Cholestasis, Extrahepatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- WallFlex Biliary Fully Covered stent (Experimental): Single arm, biliary stenting, using WallFlex Biliary Fully Covered stent
  Interventions: Device: WallFlex™ Biliary Fully Covered Metal Stent placement

INTERVENTIONS:
Device: WallFlex™ Biliary Fully Covered Metal Stent placement — Implantable metal biliary stent intended for use in the palliative treatment of biliary strictures produced by malignant neoplasms. The stent is fully covered with a polymer to reduce the potential for tumor ingrowth into the stent.

SUMMARY:
The overall objective of this study is to assess the functionality of the WallFlex™ Biliary Fully-covered stent as a palliative treatment for malignant bile duct obstruction.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Clinical symptoms of biliary obstruction
* Inoperable extrahepatic biliary obstruction by any malignant process
* Willing and able to comply with the study procedures and provide written informed consent to participate in the study.

Exclusion Criteria:

* Participation in an Investigational Study within 90 days prior to date of patient consent
* Strictures that cannot be dilated enough to pass the delivery system
* Perforation of any duct within the biliary tree
* Presence of a metal biliary stent
* Presence of any esophageal or duodenal stent
* Patients for whom endoscopic procedures are contraindicated
* Patients with known sensitivity to any components of the stent or delivery system
* Patients with active hepatitis or intrahepatic metastases that extensively involves both lobes of the liver
* Patients with an anticipated life expectancy of < 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2007-03; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bret Petersen, MD, Principal Investigator — Mayo Clinic, Rochester, MN
Locations (10):
- United States (10):
  - California Pacific Medical Center, San Francisco, California
  - Univ. of Colorado Health Sciences, Aurora, Colorado
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Duke University Med Center, Durham, North Carolina
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas
  - Univ. of VA Medical Center, Charlottesville, Virginia
  - Virginia Mason Seattle Main Clinic, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment complete
Period: Overall Study
Arm/Group | WallFlex Biliary Fully Covered Stent
Started | 74 (74 enrolled patients(signed an Informed Consent Form)were screened.58 were eligible(intent to treat))
Completed | 55 (55 out of 58 patients were evaluable(had a stent placed and had at least 1 week of follow up))
Not Completed | 19
Not completed — screen fail | 14
Not completed — Treated and later found to be ineligible | 2
Not completed — Death | 2
Not completed — Failure to deploy stent | 1

BASELINE CHARACTERISTICS:
Arm/Group | WallFlex Biliary Fully Covered Stent
Number analyzed (Participants) | 58
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 38
Age Continuous [Mean (Standard Deviation); unit: years] | 67.91 (14.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 30
Region of Enrollment [Number; unit: participants]
  United States | 58

OUTCOME MEASURES:

1. Primary Outcome: Adequate Clinical Palliation of the Biliary Obstruction
Description: Adequate clinical palliation of the biliary obstruction as demonstrated by the absence of stent occlusion within 6 month follow up or prior to death, whichever comes first in the evaluable subject cohort of 55 patients.
Time Frame: 6 months
Population: Per protocol, assessment of the primary endpoint was performed on the evaluable cohort, defined as group of patients who signed the Informed Consent Form, met eligibility criteria, received a stent and had at least one week of follow up.
Measure: Number; unit: participants
Arm/Group | WallFlex Biliary Fully Covered Stent
Number analyzed (Participants) | 55
participants | 54

2. Secondary Outcome: Technical Success
Description: Technical success is defined as the ability to deploy the stent in satisfactory position across the stricture. It was assessed in the intent-to-treat cohort.
Time Frame: At treatment
Population: Device Safety and Technical Success were evaluated for the 58 intent-to-treat patients
Measure: Number; unit: participants
Arm/Group | WallFlex Biliary Fully Covered Stent
Number analyzed (Participants) | 58
participants | 57

3. Secondary Outcome: Ability to Successfully Remove a Stent Upon Removal Attempt
Description: The ability to successfully remove a stent upon a removal attempt was defined as removal without any clinically-significant complications or technical difficulties.
Time Frame: 6 months
Population: 2 patients of the evaluable cohort (n=55) were assessed for success of stent removal without any complications/technical difficulties.
Measure: Number; unit: Participants
Arm/Group | WallFlex Biliary Fully Covered Stent
Number analyzed (Participants) | 2
Participants | 2

4. Secondary Outcome: Re-interventions
Description: Per the study protocol, re-intervention was defined as any type of endoscopic, percutaneous, or surgical procedure to improve biliary drainage after insertion of the initial stent.
Time Frame: Until 6 months or death
Population: The re-intervention rate was assessed in the evaluable cohort of 55 patients.
Measure: Number; unit: Participant
Arm/Group | WallFlex Biliary Fully Covered Stent
Number analyzed (Participants) | 55
Participant | 1

5. Secondary Outcome: Clinical Success at 1 Month After Stent Procedure as Defined by Reduction of Biliary Obstruction Symptoms
Description: Clinical success was defined as the reduction of biliary obstruction symptoms after treatment with the device.Symptoms included jaundice,pruritis,right upper quadrant abdominal pain,nausea,vomiting,fever and dark urine.For each patient,a total number of symptoms at baseline and at all post-treatment visits were recorded.Reduction in obstruction symptoms was defined as having a lower total number of symptoms at a post-treatment follow up visit compared to baseline.Here we report the number of subjects with a reduced total number of biliary obstructive symptoms at 1 month after stent treatment.
Time Frame: 1 Month
Population: 49 out of 55 evaluable subjects reached the 1-Month Follow Up visit and were evaluated for reduction of biliary obstruction symptoms.
Measure: Number; unit: Participants
Arm/Group | WallFlex Biliary Fully Covered Stent
Number analyzed (Participants) | 49
Participants | 45

6. Secondary Outcome: Clinical Success at 3 Months After Stent Procedure as Defined by the Reduction of Biliary Obstruction Symptoms
Description: Clinical success was defined as the reduction of biliary obstruction symptoms after treatment with the device.Symptoms included jaundice,pruritis,right upper quadrant abdominal pain,nausea,vomiting,fever and dark urine.For each patient,a total number of symptoms at baseline and at all post-treatment visits were recorded.Reduction in obstruction symptoms was defined as having a lower total number of symptoms at a post-treatment follow up visit compared to baseline.Here we report the number of subjects with a reduced total number of biliary obstructive symptoms at 3 months after stent treatment.
Time Frame: 3 months
Population: 34 out of 55 evaluable subjects reached the 3-Month Follow Up visit and were evaluated for reduction of biliary obstruction symptoms compared to baseline.
Measure: Number; unit: Participants
Arm/Group | WallFlex Biliary Fully Covered Stent
Number analyzed (Participants) | 34
Participants | 33

7. Secondary Outcome: Clinical Success at 6 Months After Stent Procedure as Defined by the Reduction of Biliary Obstruction Symptoms
Description: Clinical success was defined as the reduction of biliary obstruction symptoms after treatment with the device.Symptoms included jaundice,pruritis,right upper quadrant abdominal pain,nausea,vomiting,fever and dark urine.For each patient,a total number of symptoms at baseline and at all post-treatment visits were recorded.Reduction in obstruction symptoms was defined as having a lower total number of symptoms at a post-treatment follow up visit compared to baseline.Here we report the number of subjects with a reduced total number of biliary obstructive symptoms at 6 months after stent treatment.
Time Frame: 6 months
Population: 23 out of 55 evaluable subjects reached the 6-Month follow up visit and were assessed for reduction of biliary obstructive symptoms compared to baseline.
Measure: Number; unit: Participants
Arm/Group | WallFlex Biliary Fully Covered Stent
Number analyzed (Participants) | 23
Participants | 23

8. Secondary Outcome: Bilirubin Level Reduction
Description: Total bilirubin levels at 1 month follow-up were compared to initial bilirubin levels. Bilirubin level reduction was defined as total bilirubin levels being below 3mg/dl, or reduced by >30% if the initial baseline value was greater than 3mg/dl.
Time Frame: 1 month
Population: 45 out of 55 evaluable patients reported a baseline and a Month 1 total bilirubin level and were therefore analyzed for bilirubin levels reduction.
Measure: Number; unit: Participants
Arm/Group | WallFlex Biliary Fully Covered Stent
Number analyzed (Participants) | 45
Participants | 44

9. Secondary Outcome: Stent Patency at 1 Month
Description: Per the protocol, stent patency was defined as lack of obstructive symptoms and/or a total bilirubin level of less than 3mg/dl. Patency evaluations at the Month 1 visit were done on those patients with both a total bilirubin level and assessment of biliary obstructive symptoms.
Time Frame: 1 month
Population: 45 out of 55 evaluable patients had both bilirubin and obstructive symptom assessment at Month 1.
Measure: Number; unit: Participants
Arm/Group | WallFlex Biliary Fully Covered Stent
Number analyzed (Participants) | 45
Participants | 44

10. Secondary Outcome: Stent Patency at 3 Months
Description: Per the protocol, stent patency was defined as lack of obstructive symptoms and/or a normal total bilirubin level. Patency evaluations at Month 3 were done on those patients with an assessment of biliary obstructive symptoms (bilirubin levels were not measured at Month 3).
Time Frame: 3 Months
Population: 34 patients reached the Month 3 follow up point and were evaluated for stent patency.
Measure: Number; unit: Participants
Arm/Group | WallFlex Biliary Fully Covered Stent
Number analyzed (Participants) | 34
Participants | 31

11. Secondary Outcome: Stent Patency at 6 Months
Description: Per the protocol, stent patency was defined as lack of obstructive symptoms and/or a normal total bilirubin level. Patency evaluations at Month 6 were done on those patients with an assessment of biliary obstructive symptoms (bilirubin levels were not measured at Month 6).
Time Frame: 6 Months
Population: 23 patients reached the Month 6 follow up point and were evaluated for stent patency.
Measure: Number; unit: Participants
Arm/Group | WallFlex Biliary Fully Covered Stent
Number analyzed (Participants) | 23
Participants | 21

12. Secondary Outcome: Time to Stent Occlusion
Description: Time to stent occlusion(measured in days since stent placement) was recorded for any subjects who experienced occlusion.
Time Frame: Until 6 Months or death
Population: Only 1 subject experienced stent occlusion during the study.
Measure: Number; unit: Days
Arm/Group | WallFlex Biliary Fully Covered Stent
Number analyzed (Participants) | 1
Days | 142

13. Secondary Outcome: Number of Device-Related Adverse Events
Description: Adverse Events reported during the trial were evaluated for their device-and procedure-relatedness and severity in order to assess device safety. An adverse event was defined as any untoward medical occurance in a study participant.
Time Frame: Until 6 months or death
Population: The intent-to-treat cohort of 58 patients was used for this analysis. Of all the events reported for this population, only 6 events were reported as device-related.
Measure: Number; unit: Events
Arm/Group | WallFlex Biliary Fully Covered Stent
Number analyzed (Participants) | 58
Events | 6

ADVERSE EVENTS:
Time Frame: 11 months
Arm/Group | WallFlex Biliary Fully Covered Stent
Serious Adverse Events (participants affected / at risk) | 45/58
Other Adverse Events (participants affected / at risk) | 38/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | WallFlex Biliary Fully Covered Stent (N=58)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3)
Abscess (Infections and infestations) | 1 (1)
Asthenia (General disorders) | 2 (2)
Bacteraemia (Infections and infestations) | 1 (1)
Cardiac Failure Congestive (Cardiac disorders) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Chest pain (General disorders) | 2 (2)
Cholangitis (Hepatobiliary disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 2 (2)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Death (General disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 4 (4)
Diverticular Perforation (Gastrointestinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Enterovesical Fistula (Gastrointestinal disorders) | 1 (1)
Gall bladder perforation (Hepatobiliary disorders) | 1 (1)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 1 (1)
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Obstruction gastric (Gastrointestinal disorders) | 1 (1)
Oedema peripheral (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Pancreatic Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 18 (18)
Pancreatic Carcinoma Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 (8)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Posprocedural hemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pyrexia (General disorders) | 3 (3)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Vomitting (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | WallFlex Biliary Fully Covered Stent (N=58)
Abdominal pain (Gastrointestinal disorders) | 6 (6)
Ascites (Gastrointestinal disorders) | 5 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5)
Constipation (Gastrointestinal disorders) | 4 (4)
Nausea (Gastrointestinal disorders) | 6 (6)
Oedema peripheral (General disorders) | 3 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pyrexia (General disorders) | 3 (3)
Vomitting (Gastrointestinal disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No